CLINICAL TRIAL: NCT01378455
Title: Effectiveness of Interactive Computerized Handwriting Training Program on Handwriting Performance in Children With Cerebral Palsy
Brief Title: Effectiveness of Handwriting Training Program on Handwriting Performance in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 98-3193B
Record Dates: First submitted 2011-06-21; First posted 2011-06-22 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2011-05

CONDITIONS: Cerebral Palsy
Keywords: handwriting; cerebral palsy; visual perception; sensory function; motor function; computerized handwriting programs
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ICHTP group (Experimental): In ICHTP (interactive computerized handwriting training program) group, they received the training of visual-perception .visual-motor integration skill of children and modulate muscle strength of grasp through ICHTP software
  Interventions: Other: interactive computerized handwriting training program
- THTP group (Active Comparator): The THTP (traditional handwriting training program)group ,they received the training of paper-pencil activities with visual-perception and visual-motor integration skills
  Interventions: Other: traditional handwriting training program

INTERVENTIONS:
Other: interactive computerized handwriting training program — In ICHTP group, they received the training of visual-perception .visual-motor integration skill of children and modulate muscle strength of grasp through ICHTP software. The training program costs 45 min/once, three times/one week, and sustains four weeks.In traditional group, they received the training of paper-pencil activities with visual-perception and visual-motor integration skills. The training duration is as long as ICHTP group.
  Other Names: computerized handwriting training program
  Arms: ICHTP group
Other: traditional handwriting training program — The THTP group ,they received the training of paper-pencil activities with visual-perception and visual-motor integration skills
  Arms: THTP group

SUMMARY:
Visual perception impairment and upper limb disability will affect the handwriting performance. Children with cerebral palsy (CP) who have good function on upper extremity may associated with visual perception impairment, which will impact the handwriting performance. However, there were few studies to investigate the handwriting problems in children with CP who have good upper limb functions. To date, there are no studies to investigate the effectiveness of computerized handwriting training programs on handwriting performance in children with CP. The aims of this study were to establish the relationships of visual perception, visual motor integration, and motor coordination of handwriting performance in children with typical development (TD) in Taiwan, to establish the norms of handwriting performance in children with TD in Taiwan, to compare handwriting performance in children with CP and children with TD, to clarify the relationship of visual perception function and handwriting performance in children with CP, and to examine the effectiveness of interactive computerized handwriting training program (ICHTP) on handwriting performance in children with CP.

The investigators will collect 90 children with TD and 48 children with CP in the 1st phase. All children will receive clinical and Chinese handwriting assessment tool (CHAT) assessments. The CHAT and ICHTP will be modified as Taiwan-version handwriting assessment tool and training programs for children in Taiwan, respectively. Clinical assessments include the visual perception, visual motor integration, fine motor skill, and handwriting performance. The CHAT assessed the handwriting legibility, accuracy, pen pressure and writing speed. In the 2nd phase, the investigators will collect 48 children with CP, who were randomly classified into ICHTP group and Traditional Handwriting Training Program (THTP). All children with CP will receive clinical and CHAT assessments before and after interventions.

The expected results of this study are the visual perception function is related to handwriting performance in children with CP, and the improvements in the handwriting legibility, accuracy, pen pressure and writing speed of ICHTP training group are greater than THTP training group.

DETAILED DESCRIPTION:
This study were to establish the relationships of visual perception, visual motor integration, and motor coordination of handwriting performance in children with TD in Taiwan, to establish the norms of handwriting performance in children with TD in Taiwan, to compare handwriting performance in children with CP and children with TD, to clarify the relationship of visual perception function and handwriting performance in children with CP in the first phase, and to examine the effectiveness of interactive computerized handwriting training program (ICHTP) via a randomized controlled study in children with CP in the second phase.The subjects are ninety children with typical development aged between 6-12 years from elementary school and forty-eight children with CP aged between 6-12 years from Chang Gung Memorial Hospital (Taipei branch, Linkou branch, Taoyuan branch, Kaohsiung branch), Far Eastern Memorial Hospital, Taipei Veterans General Hospital and Buddhist Tzu Chi General Hospital (Taipei branch)etc.Experimental design In first phase, we establish the relationships of visual perception, visual motor integration, and motor coordination of handwriting performance in children with TD in Taiwan, to establish the norms of handwriting performance in children with TD among different age groups in Taiwan, a comparison designed study to compare the handwriting performance among 2 CP groups and TD groups. All children were assigned into diplegia group, hemiplegia group, and typical development (TD) group. Then we will assessment the fine motor skill, visual perception and handwriting performance by occupational therapist.

Experimental procedures:

All children were assessed with clinical assessments and the Chinese handwriting assessment tool (CHAT). Clinical assessments included Manual Ability Classification System (MACS), Bruininks-Oseretsky Test of Motor Proficiency-second edition (BOT-II), the Test of Visual-Perceptual Skills Revised (TVPS-R), Beery-Buktenica Developmental Test of Visual-Motor Integration (Berry VMI) and comprehensive test of basic reading and writing. Evaluations were performed in about 1.5-2 hours in a silent and restful room, eliminating factors such as fatigue and distraction of attention and concentration, which could have an impact on the results. All the tests used in the study were individually administered to all children. The performance of all children was videotaped for later scoring.

In second phase, all CP children were randomized assigned into ICHTP group or THTP group. All participations will received clinical and CHAT assessments before and after intervention. Clinical assessments included Manual Ability Classification System (MACS), Bruininks-Oseretsky Test of Motor Proficiency-second edition (BOT-II), the Test of Visual-Perceptual Skills Revised (TVPS-R), Beery-Buktenica Developmental Test of Visual-Motor Integration (Berry VMI) and comprehensive test of basic reading and writing. Evaluations were performed in about 2 hours in a silent and restful room, eliminating factors such as fatigue and distraction of attention and concentration, which could have an impact on the results. All the tests used in the study were individually administered to all children. The performance of all children was videotaped for later scoring. The intervention consisted of ICHTP and THTP training programs, which is 45 min/once, three times/one week, and sustain four weeks.

ELIGIBILITY:
Inclusion Criteria:

* ability to follow instructions and complete the assessment
* agreement to join this study.
* CP with hemiplegia and diplegia
* Manual Ability Classification System (MACS) of dominant hand: levels 1-2

Exclusion Criteria:

* psychosocial, behavioral and emotional problems, such as ADHD, and autism.
* physical dysfunction, such as neuromuscular disorders.
* significant hearing or visual impairment
* significant sensory impairment.
* Learning disability
* Test of Nonverbal Intelligence( TONI-2) less than two standard deviation,
* unstable medical situation (ex: seizure).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Body function and structure | pre-treatment, post-treatment, 3 months, 6 months, 12 months
  pre-treatment, post-treatment, 3 months, 6 months, 12 months Body function and structure: TVPS, Reading and handwriting tests, SP, etc.

SECONDARY OUTCOMES:
Activities and participation | pre-treatment, post-treatment, 3 months, 6 months, 12 months
  pre-treatment, post-treatment, 3 months, 6 months, 12 months
  Activities and participation: SFA,CAPE, PAC, etc.
Quality of life | pre-treatment, post-treatment, 3 months, 6 months, 12 months
  pre-treatment, post-treatment, 3 months, 6 months, 12 months HRQOL: CPQOL, etc.
Computer Analysis for Chinese Handwriting(CACH) | pre-treatment, post-treatment, 3 months, 6 months, 12 months
  pre-treatment, post-treatment, 3 months, 6 months, 12 months
  Computer Analysis for Chinese Handwriting(CACH)

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling Chen, MD,PhD, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taoyuan, Taiwan